CLINICAL TRIAL: NCT01216514
Title: Differential Characteristics of All Serologic Markers for Chronic Inflammatory Bowel Diseases During Clinical Forms With Weak or Strong Evolution Capacities
Brief Title: Serologic Markers for Inflammatory Bowel Disease During Clinical Forms With Weak or Strong Evolution Capacities
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1008074
Record Dates: First submitted 2010-10-04; First posted 2010-10-07 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-11

CONDITIONS: Inflammatory Bowel Diseases
Keywords: chronic inflammatory bowel diseases; crohn disease; hemorrhagic rectocolitis; immunological markers; serological markers; ANCA; ASCA
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Proctocolitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Factors forecast Chronic Inflammatory Bowel Diseases (IBD) remain at present essentially on clinical factors (extension of the disease, achievement of the perianal ring, requirement of surgery, treatment by immunomodulators…). All IBD specific immunological or serological markers showed only a diagnostic role for indefinite colitis (hemorrhagic Rectocolitis vs Crohn Disease) but were never able to be considered as predictive elements of adults IBD evolution. Among the most used, the presence of ANCA's antibody and ASCA allows to separate hemorrhagic rectocolitis (ANCA + / ASCA-) from Crohn disease (ANCA-/ASCA +) and their combination present an average sensibility about 85 % and a 85 % specificity. However, 8 other antibody types were recently isolated and estimated individually during IBD in particular during child Crohn diseases (anti-OmpC, anti-I2, anti-CBir1, anti-glycans (ALCA, AMCA and ACCA) anti-Goblet cells and albicans Candida's specific anti-mannan). These complementary assays improve significantly the reliability of the diagnosis. However, if the use of these new markers has an indisputable diagnostic role, their predictive role in the evolution of IBD was estimated at the adult's only rarely during Crohn diseases. Consequently, the investigators suggest realizing an exhaustive analysis of all these new immunological markers to define, if their association can have an interest in the differentiation of stable (or little evolutionary) and unstable (or quickly evolutionary) clinical forms.

ELIGIBILITY:
Inclusion Criteria:

* Major Patient
* IBD (RCH or MC) diagnosed according to the clinical, endoscopic and histological criteria
* Accepting the sampling of blood
* Patient member or legal successor of a national insurance scheme
* Taken care medical in the service of gastroenterology of CHU de Saint Etienne
* Patient having signed the form of consent

Exclusion Criteria:

* Minor Patient or uncapable
* Patient suffering from indefinite colitis
* Refusal of the sampling of blood
* Pregnant Woman
* Incapacity or refusal to sign the consent writes
* Subjects deprived of freedom by a court or administrative order
* Use of an anti-TNF. According to the indications ensuing from the Sonic trial or from the strategy " Top Down ".

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
definition of the unstable form of Crohn disease and RCH | day 1
  Crohn disease, at least one of the following criteria:
  Use of anti-TNF antibody in case of immunosuppressor failure. Surgery of resection (at least two resections or more than 70 cms of intestinal resections) Anoperineal form with complex fistulas Spread intestinal affection Beginning of the disease before 16 years
  RCH, at least one of the following criteria:
  Initial pancolite affection Immunosuppresseur use in the first year of evolution Use of anti-TNF Severe Colitis

SECONDARY OUTCOMES:
Treatment effective : patient in clinical and endoscopic remission state | day 1
  Treatment will be considered as effective if the patient is in clinical and endoscopic remission state.
  A patient will be considered in clinical remission if he presents:
  * A CDAI score (Crohn disease activity index) lower than 150 for the MC;
  * A MAYO score lower than 2 or a score of Lichtiger lower than 4 for RCH.
  A patient will be considered in endoscopic remission if he presents:
  * A Lichtiger score lower than 4 for the MC;
  * An endoscopic MAYO score lower than 2 for RCH.
corticodependant patient | history and day 1
  A patient will be considered as corticodependant if he presents a push of IBD after decresase of the corticosteroid therapy on 2 occasions.
corticoresistant patient | history and day 1
  A patient will be considered as corticoresistant if his disease remains active for a threshold of corticosteroid therapy of at least 40 mg/day of Prednisolone and on a duration of 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: ROBLIN Xavier, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- Service de Gastro-entérologie, Saint-Etienne, France